CLINICAL TRIAL: NCT02282319
Title: Influence of Spinal or Intravenous Dexmedetomidine on Spinal Anesthesia With Chloroprocaine and Bladder Function in Day-case Surgery. A Double Blind Randomized Study.
Brief Title: Spinal or Intravenous Dexmedetomidine in Ambulatory Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Dr M. B. Breebaart, dr, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 13/35/334
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Surgery Ambulatory
Keywords: spinal or intravenous dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A chloro (Experimental): spinal chloroprocaine 40 mg
  Interventions: Other: spinal chloroprocaine 40 mg
- B chloro+ spin dexdor (Experimental): Spinal chloroprocaine 40 mg spinal dexmedetomidine 0.5 mcg
  Interventions: Drug: spinal dexmedetomidine 0.5 mcg; Other: spinal chloroprocaine 40 mg
- C chloro + IV dexdor (Experimental): Spinal chloroprocaine 40 mg IV dexmedetomidine 0.5 mcg/kg
  Interventions: Other: spinal chloroprocaine 40 mg; Drug: IV dexmedetomidine 0.5 mcg/kg

INTERVENTIONS:
Drug: spinal dexmedetomidine 0.5 mcg — Administration of dexmedetomidine 0.5 mcg
  Other Names: dexdor
  Arms: B chloro+ spin dexdor
Other: spinal chloroprocaine 40 mg — spinal anesthesia with chloroprocaine 40 mg
  Other Names: ampres
Drug: IV dexmedetomidine 0.5 mcg/kg — intravenous administration of dexmedetomidine 0.5 mcg/kg
  Other Names: dexdor
  Arms: C chloro + IV dexdor

SUMMARY:
The primary objective of this double blind randomized study is to determine the effect of dexmedetomidine on onset and duration of the sensory and motor block and on the influence on bladder function after spinal anesthesia with chloroprocaine. Our primary hypothesis is that sensory block will significantly be prolonged by dexmedetomidine administered by both the spinal and the intravenous route. The investigators do not expect a significant difference in motor block duration between intravenous or spinal administration. Secondary outcomes are micturition problems, duration of analgesia and the occurrence of side effects such as sedation and hypotension.

DETAILED DESCRIPTION:
The study is designed as a multicenter study and randomization and inclusion of patients will be performed in three hospitals. Each hospital has its own randomisation sequence and coordinating investigator who will be responsible for appointing blinded and unblinded participators in the study.

Patients scheduled for spinal anesthesia in ambulatory surgery will be randomized by sealed envelopes (computer generated sequence) into one of the following three study groups:

spinal chloroprocaine 40 mg with spinal dexmedetomidine (5mcg) spinal chloroprocaine 40 mg with intravenous dexmedetomidine ( 0.5 mcg/kg) spinal chloroprocaine 40 mg alone (control group)

All patients will receive the same amount of spinal solution, containing chloroprocaine 1% (4 ml) with dexmedetomidine (0.5 ml, 1 mcg/ml) or NaCl ( sodiumchloride) 0,9% (0.5 ml ) ( and 50 ml intravenous Nacl 0.9, containing dexmedetomidine (0.5 mcg/kg) or not depending on the study group. All solutions are prepared by an independent anesthesiologist and labelled as Intravenous study medication and spinal study medication. Spinal anesthesia and data registration will be done by a blinded anesthesist and/or study nurse on a data sheet designed for the study.

Spinal anesthesia is performed in the lateral decubitus at L3-L4 vertebral interspace and standard monitoring for this procedure is applied. Insufficient analgesia will be treated with sufentanil increments. Hypotension and bradycardia will be treated with ephedrine and atropine. Patients will be discharged when the block is regressed, there is no sedation or nausea and nrs scores of pain are below 4. Patients will be contacted by telephone after one week to evaluate any postoperative complaints.Micturition will receive a score based on bladder volumes measured by bladder scanning and subjective complaints . This score system was used in two of our former studies (1,2)

To calculate the power of this study, we used the mean L2 regression of a previous study after spinal chloroprocaine with its standard deviation (SD 20 min, mean 90 min) and compared it to a mean increase with 30 %. We calculated that we should include 7 patients in each group to obtain a power of 80%.

To be sure to detect a possible difference in discharge time as well, we calculated a sample size of 48 patients for each group to detect a 30-minute difference.

Statistical analysis will be done with ANOVA analysis , A kruskal-Wallis of Mann Whitney test depending on the distribution of the population and if the values are parametric or not. This will be done by spss.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) class 1 & 2,
* undergoing day-case knee arthroscopy

Exclusion Criteria:

* micturition problems,
* neurological history or
* previous lower abdominal surgery with an abnormal micturition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
sensory block regression L2 dermatome (minutes) (Time from injection until First time registration of loss of cold sensation) | up to 360 minutes
  Time from injection until First time registration of loss of cold sensation at the L2 dermatome during block regression. Loss of cold sensation will be regularly assessed from spinal injection until total regression of the sensory block
Motor block regression (minutes) (time from injection until achievement of active knee movement) | up to 240 minutes
  time from injection until achievement of active knee movement during block regression. Motor block will be assessed at regular intervals from spinal injection untill total regression of the motor block

SECONDARY OUTCOMES:
discharge time (minutes) | up to 240 minutes
  time from spinal injection until achievement of discharge criteria
time to micturition ( minutes) | up to 240 minutes
  time from injection until first voiding
blood pressure drop | up to 240 minutes
  percentage of drop blood pressure compared to base line ( measured before spinal injection) . Blood pressure will be measured at regular intervals from just prior to spinal injection until discharge

OTHER OUTCOMES:
micturition problems (scaling based on bladder volumes and subjective difficulties) in a 1-5 point scale | at discharge ( up to 240 minutes)
  classification of problems ( scaling based on bladder volumes and subjective difficulties) in a 1-5 point scale

CONTACTS AND LOCATIONS:
Overall Officials: margaretha breebaart, MD, Principal Investigator — University Hospital, Antwerp; Marcel Vercauteren, MD, PHD, Principal Investigator — University Hospital, Antwerp
Locations (2):
- Belgium (2):
  - University Hospital Antwerp, Antwerp
  - Sint Augustinus, Wilrijk

REFERENCES:
- [Background] Breebaart MB, Vercauteren MP, Hoffmann VL, Adriaensen HA. Urinary bladder scanning after day-case arthroscopy under spinal anaesthesia: comparison between lidocaine, ropivacaine, and levobupivacaine. Br J Anaesth. 2003 Mar;90(3):309-13. doi: 10.1093/bja/aeg078. PMID 12594142
- [Background] Breebaart MB, Teune A, Sermeus LA, Vercauteren MP. Intrathecal chloroprocaine vs. lidocaine in day-case surgery: recovery, discharge and effect of pre-hydration on micturition. Acta Anaesthesiol Scand. 2014 Feb;58(2):206-13. doi: 10.1111/aas.12247. PMID 24563922